CLINICAL TRIAL: NCT06867133
Title: The Evaluation of the Curative Effect of Electrophysiological Rehabilitation Services on Endometrial Repair After Induced Abortion
Acronym: rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ChiCTR2400091098
Record Dates: First submitted 2025-02-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Endometrium
Keywords: endometrium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrophysiological Rehabilitation Group (Experimental): On the basis of treatment in the control group, postoperative electrophysiological rehabilitation services were started for 30 minutes each time, once a day, for 6 consecutive days as one course of treatment, for a total of one course of treatment. The patch is located at the projection site of the lower abdomen uterus as shown in the figure, simulating bioelectric stimulation parameters: biphasic pulse current, frequency 2Hz, pulse width 3ms.
  Simultaneously conducting family health education, including but not limited to:
  1. Guidance on postoperative physical recovery after abortion: provide advice on postoperative care, nutrition, activity, and personal hygiene;
  2. Introduction to contraceptive methods: Introduce the advantages and disadvantages of various contraceptive methods, and help patients choose the most suitable contraceptive method for themselves;
  3. Other related health education: including fertility planning and the best time to conceive again.
  Interventions: Device: Electrophysiological rehabilitation
- control group (No Intervention): Accept routine health education and follow-up after induced abortion surgery, excluding specialized home health education services and biomimetic electrical stimulation therapy. Pay attention to postoperative recovery, usually through telephone or outpatient follow-up, and receive routine anti infective treatment after surgery.

INTERVENTIONS:
Device: Electrophysiological rehabilitation — On the basis of treatment in the control group, postoperative electrophysiological rehabilitation services were started for 30 minutes each time, once a day, for 6 consecutive days as one course of treatment, for a total of one course of treatment. The patch is located at the projection site of the lower abdomen uterus as shown in the figure, simulating bioelectric stimulation parameters: biphasic pulse current, frequency 2Hz, pulse width 3ms.
  Simultaneously conducting family health education, including but not limited to:
  1. Guidance on postoperative physical recovery after abortion: provide advice on postoperative care, nutrition, activity, and personal hygiene;
  2. Introduction to contraceptive methods: Introduce the advantages and disadvantages of various contraceptive methods, and help patients choose the most suitable contraceptive method for themselves;
  3. Other related health education: including fertility planning and the best time to conceive again.
  Arms: Electrophysiological Rehabilitation Group

SUMMARY:
Exploring the efficacy evaluation of electrophysiological rehabilitation services in endometrial repair after induced abortion, providing scientific basis for medical institutions and government post abortion care decision-making.

This study is a multicenter randomized controlled intervention study. The main endpoint of the study was the measurement of endometrial thickness by transvaginal ultrasound on days 21-23 after abortion.

Secondary study endpoint:

1. Postoperative uterine contraction pain;
2. Patient satisfaction;
3. Menstrual recurrence time;
4. Changes in menstrual flow for two consecutive periods after surgery;
5. The duration of two consecutive menstrual periods after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18-40 years old;
2. Previous menstrual patterns;
3. Pregnancy duration 6-10 weeks;
4. Ultrasound indicates intrauterine pregnancy;
5. Voluntarily accepting surgical induced abortion with no contraindications for induced abortion;
6. Voluntarily participate in the trial and sign the informed consent form.
7. Patients or their families are able to understand the research protocol and are willing to participate in this study, providing written informed consent.

Exclusion Criteria:

1. Medical abortion patients;
2. Patients with pelvic and abdominal benign and malignant tumors and other systemic diseases; C) Skin problems such as ulceration, infection, and blisters at the treatment site;

d) Patients with missed miscarriage diagnosed clinically; e) Patients with combined uterine fibroids, adenomyosis, and uterine malformations; f) Those who have inserted intrauterine devices (including copper containing intrauterine devices and levonorgestrel containing intrauterine devices); g) Individuals who have had three or more previous induced abortions; h) Clinical diagnosis of thin endometrium; i) Individuals with a history of cesarean section surgery; j) Individuals with severe mental illnesses; k) Researchers determine other situations that are not suitable for participating in this study; l) Patients or their families are unable to understand the conditions and objectives of this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Transvaginal ultrasound examination is used to measure the thickness of the endometrium. | On the 21st to 23rd day after abortion.
  On the 21st to 23rd day after abortion, vaginal ultrasound was used to measure endometrial thickness.

SECONDARY OUTCOMES:
Postoperative uterine contraction pain | One week after surgery
  The degree of postoperative pain was evaluated using the Visual Analogue Scale (VAS) scoring method. A horizontal line of 10 cm in length was drawn, with the two ends representing 0 and 10 respectively. 0 indicated no pain, and 10 represented the most unbearable pain that could be imagined. Patients were asked to select the corresponding number based on their postoperative pain sensation to describe the intensity of their subjective pain. The time for postoperative pain assessment was as follows: for the experimental group, the VAS pain score was evaluated before treatment on the second day after surgery and after one session of bioelectrical stimulation treatment; for the control group, the VAS pain score was evaluated only once on the second day after surgery.
Patient satisfaction | 3 months after surgery
  Survey the satisfaction levels of patients in the control group and intervention group, specifically covering sub item satisfaction evaluations of biomimetic electrical stimulation treatment, doctor attitude, abortion process, and extended home rehabilitation services. Each item is divided into five levels: very satisfied, satisfied, average, dissatisfied, and very dissatisfied. In addition, the overall satisfaction of the above four items will be comprehensively evaluated.
Menstrual recurrence time | 3 months after surgery
  Observe the time of menstrual recurrence in two groups after surgery, that is, the interval between the completion of induced abortion and the recurrence of menstruation in the subjects.
Changes in menstrual flow for two consecutive periods after surgery | 3 months after surgery
  Understand the postoperative menstrual flow of the research subjects for two consecutive periods. The specific reference criteria are: compared with the preoperative menstrual flow, it is divided into five levels: much more, slightly more, similar, slightly less, and much less.
Duration of two consecutive menstrual periods after surgery | 3 months after surgery
  By conducting a 3-month online follow-up on the control group and intervention group, we aim to understand the duration of continuous menstruation in the study subjects after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR